CLINICAL TRIAL: NCT01797588
Title: Pain After Total Knee Arthroplasty: A Randomized Controlled Trial Examining the Effectiveness of a Combined Adductor-canal Peripheral Nerve Block With Periarticular Infiltration Versus Adductor-canal Nerve Block Alone Versus Periarticular Infiltration Alone.
Brief Title: Pain After Total Knee Arthroplasty: A Trial Examining Combined Adductor-canal Nerve Block and Periarticular Infiltration Versus Adductor Canal Nerve Block Versus Periarticular Infiltration
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: North York General Hospital (Other)
Responsible Party: Principal Investigator, Mona Sawhney, Dr. Mona Sawhney, NP, North York General Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: NYGHTKA-01
Record Dates: First submitted 2013-02-20; First posted 2013-02-22 (Estimated); Last update posted 2015-01-05 (Estimated); Status verified 2015-01

CONDITIONS: Total Knee Arthroplasty; Postoperative Pain
Keywords: Total Knee Arthroplasty; Pain; Periarticular infiltration; Adductor canal block; Postoperative
MeSH Terms: conditions — Pain, Postoperative; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- adductor-canal block and periarticular infiltration (Active Comparator): Adductor-canal block,performed prior to surgery using ultra sound guidance by an anesthetist, with a total of 30mL of 0.33% ropivacaine injected into the area surrounding the saphenous nerve. Periarticular infiltration, performed intra-operatively by the surgeon, involves administering a 110 mL solution of ropivacaine 300mg, preservative free morphine 10mg, ketorolac 30mg mixed in normal saline into the knee.
  Interventions: Procedure: Adductor-canal block; Procedure: Periarticular infiltration
- adductor-canal block (Active Comparator): The adductor-canal block only group will receive an adductor-canal block prior to surgery in the block room using ultra sound guidance by an anesthetist. After the adductor-canal is located a total of 30mL of 0.33% ropivacaine will be injected into the area surrounding the saphenous nerve. Participants will also receive 110mL of normal saline administered as follows: the first 20mL aliquot is injected into the posterior capsule and the medial and lateral ligaments just prior to implantation; after the implants have been cemented and curing, another 20mL is infiltrated to the quadriceps and retinacular tissues. The remaining solution (~60mL) is used to infiltrate the muscle, subcutaneous tissues.
  Interventions: Procedure: Adductor-canal block
- periarticular infusion group (Active Comparator): Periarticular infiltration,performed intra-operatively,involves administering a 110 mL solution of ropivacaine 300mg, preservative free morphine 10mg, ketorolac 30mg mixed in normal saline into the knee. It will be administered as follows: the first 20mL aliquot is injected into the posterior capsule and the medial and lateral ligaments just prior to implantation; after the implants have been cemented and curing, another 20mL is infiltrated to the quadriceps and retinacular tissues. The remaining solution (~60mL) is used to infiltrate the muscle, subcutaneous tissues.
  Interventions: Procedure: Periarticular infiltration

INTERVENTIONS:
Procedure: Adductor-canal block — The adductor-canal will be located via ultra sound and a total of 30mL of 0.33% ropivacaine will be injected into the area surrounding the saphenous nerve.
  Arms: adductor-canal block; adductor-canal block and periarticular infiltration
Procedure: Periarticular infiltration — Periarticular infiltration will be performed intra-operatively and involves administering a 110 mL solution of ropivacaine 300mg, preservative free morphine 10mg, ketorolac 30mg mixed in normal saline into the knee. In each Knee: the first 20mL aliquot is injected into the posterior capsule and the medial and lateral ligaments just prior to implantation; after the implants have been cemented and curing, another 20mL is infiltrated to the quadriceps and retinacular tissues. The remaining solution (~60mL) is used to infiltrate the muscle, subcutaneous tissues.
  Arms: adductor-canal block and periarticular infiltration; periarticular infusion group

SUMMARY:
Effective pain management following total knee arthroplasty is important to facilitate early mobilization and rehabilitation. To manage post-operative pain, multimodal analgesia, including acetaminophen, NSAID's, gabapentin, opioids and local anesthetics are used. However, local anesthetics injected into the femoral nerve area may cause a block in motor function of the quadriceps muscle. Both adductor-canal peripheral nerve block performed pre-operatively, and periarticular infiltration performed intra-operatively are effective in reducing pain following TKA without causing quadriceps motor block which can impede mobilization. No published trials have been found that compare single shot adductor-canal block plus periarticular infiltration to periarticular infiltration only or adductor-canal nerve block only. The purpose of this trial is to examine the effect of 3 different approaches to nerve blockade: 1) adductor-canal block plus periarticular infiltration; 2) adductor-canal block only; 3) periarticular infiltration only, on pain, analgesic consumption, mobility, pain related interference with activities and length of hospital stay in participants undergoing unilateral TKA. Patients will be eligible for participation if they are 18 years old or older, and can speak, and read English. Ninety-six trial participants will be randomized to receive 1 of the 3 approaches to nerve blockade as part of their pain management plan. Outcomes will be measured on post-operative days 1 and 2 and length of stay will be calculated in hours after the participant is discharged to home. It is hypothesized that participants that receive both adductor-canal nerve block plus periarticular infiltration will report less pain, improved mobility and less pain related interference with activities.

DETAILED DESCRIPTION:
Hypothesis:

The combination of adductor-canal peripheral nerve block with periarticular intra-operative infiltration (AC+PI) provides superior analgesia and preserves motor function as compared to adductor-canal block (AC) only or periarticular infusion (PI) only.

Specific Aims:

The primary outcome of this trial is to examine pain on walking, using a 0 to 10 numeric rating scale (NRS), at post-operative day 1 in patients who undergo TKA using 3 different approaches to nerve blockade: 1) adductor-canal block plus periarticular infiltration; 2) adductor-canal block only; 3) periarticular infiltration only.

The secondary outcomes of this trial are to examine, in patients who undergo TKA using 3 different approaches to nerve blockade: 1) adductor-canal block plus periarticular infiltration; 2) adductor-canal block only; 3) periarticular infiltration only:

1. pain at rest on post-operative day 1 and day 2 at 1000
2. pain with walking on post-operative day 2
3. pain with knee flexion on post-operative day 1 and day 2 at 1000
4. analgesic consumption on post-operative day 1 and day 2
5. distance walked on post-operative day 1 and day 2
6. pain related interference with activities on post-operative day 1 and day 2
7. length of stay

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older
* ASA I-III
* eligible for spinal anesthetic
* able to speak
* read and understand English
* willing to participate in the trial
* will be discharged home.

Exclusion Criteria:

* contraindication to regional anesthesia
* have an allergy to local anesthetics
* contradiction to NSAID's
* have chronic pain that is not related to their knee joint
* have been using opioids on a chronic basis (3 months or longer)
* have a pre-existing peripheral neuropathy involving the operative site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2013-03; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | Post-operative day 1
  The primary outcome of this trial is to examine pain on walking, using a 0 to 10 numeric rating scale (NRS), at post-operative day 1 in patients who undergo TKA

SECONDARY OUTCOMES:
pain related interference with activities | on post-operative day 1 and day 2
  This will be measured using the BPI-interference subscale.

CONTACTS AND LOCATIONS:
Overall Officials: Monakshi Sawhney, PhD, Principal Investigator — North York General Hospital
Locations (1):
- North York General Hospital, Toronto, Ontario, Canada